CLINICAL TRIAL: NCT00997139
Title: Clearance of Nasal Staphylococcus Aureus Colonization With Triple Antibiotic Ointment
Brief Title: Clearance of Nasal Staphylococcus Aureus With Triple Antibiotic Ointment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dennis West, Professor in Dermatology and Pediatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU-9892
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Nasal Carriers of Staphylococcus Aureus
Keywords: healthcare; staphylococcus aureus; nasal
MeSH Terms: conditions — Staphylococcal Infections | interventions — bacitracin zinc, neomycin sulfate, polymyxin B, drug combination; Neomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Neosporin (polymyxin B 5,000units, bacitracin 400 units, neomycin 3.5mg) — 2 1/32oz packages will be dispensed. If positive nasal swab for S. aureus, subjects will apply a small amount to anterior nares twice daily for 5 days.

SUMMARY:
Staphylococcus aureus, a bacteria that lives commonly in the anterior nostrils, is seen in about 30% of healthcare workers. Applying mupirocin ointment, a prescription, to the nostrils twice daily for 5 days is the current standard of care for treatment to clear this bacteria. This research study is designed to determine the rate of clearance of this bacteria in healthcare workers who are carriers when using triple antibiotic ointment instead of mupirocin ointment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Must have consented prior to registration for the study

Exclusion Criteria:

* active infection
* concurrent treatment with antibiotics, topical or systemic
* S. aureus decolonization attempt in prior six months
* history of HIV
* chemotherapy or systemic immunosuppressive therapy
* history of neomycin allergy or sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lio, MD, Principal Investigator — Northwestern Unviersity
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only subjects with a positive Baseline culture continued on a treatment arm.
Period: Overall Study
Arm/Group | All Subjects
Started | 216
Treated for Positive Baseline Culture | 30
Completed | 30
Not Completed | 186

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Baseline culture positive for Staphylococcus aureus
Arm/Group | Treatment Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Carrier Rate for Staphylococcus Aureus
Description: Percentage of subjects with baseline culture positive for Staphylococcus aureus (via nasal swab)
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Groups:
- All Subjects: All subjects enrolled
Arm/Group | All Subjects
Number analyzed (Participants) | 216
percentage of subjects | 20.8

2. Primary Outcome: MSSA Clearance Rate
Description: Percentage of subjects with methicillin-sensitive S. aureus on Baseline culture who achieved clearance with treatment.
Time Frame: 14 days
Measure: Number; unit: percentage of subjects
Groups:
- MSSA: Baseline culture positive for methicillin-susceptible staphylococcus aureus
Arm/Group | MSSA
Number analyzed (Participants) | 28
percentage of subjects | 57.1

3. Primary Outcome: MRSA Clearance Rate
Description: Percentage of subjects with methicillin-resistant S. aureus on Baseline culture who achieved clearance with treatment.
Time Frame: 14 days
Measure: Number; unit: percentage of subjects
Groups:
- MRSA: Subjects with Baseline culture positive for methicillin-resistant Staphylococcus aureus
Arm/Group | MRSA
Number analyzed (Participants) | 2
percentage of subjects | 0

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/216
Other Adverse Events (participants affected / at risk) | 0/216

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes